CLINICAL TRIAL: NCT02493335
Title: Double-blind, Randomized, Placebo-controlled, Phase III Study on the Efficacy and Tolerability of a 48-week Treatment With Two Different Doses of Budesonide Effervescent Tablets vs. Placebo for Maintenance of Clinico-pathological Remission in Adult Patients With Eosinophilic Esophagitis
Brief Title: Maintenance of Remission With Budesonide Orodispersible Tablets vs. Placebo in Eosinophilic Esophagitis
Acronym: EOS-2
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Dr. Falk Pharma GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BUL-2/EER; 2014-001485-99 (EudraCT Number)
Record Dates: First submitted 2015-07-07; First posted 2015-07-09 (Estimated); Last update posted 2021-10-07 (Actual); Status verified 2021-10

CONDITIONS: Eosinophilic Esophagitis
MeSH Terms: conditions — Eosinophilic Esophagitis | interventions — Budesonide; BID protein, human

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Budesonide 0.5mg orodispersible tablet twice daily (Experimental): Budesonide 0.5mg orodispersible tablet twice daily
  Interventions: Drug: Budesonide 0.5mg orodispersible tablet twice daily
- Budesonide 1mg orodispersible tablet twice daily (Experimental): Budesonide 1mg orodispersible tablet twice daily
  Interventions: Drug: Budesonide 1mg orodispersible tablet twice daily
- Placebo orodispersible tablet twice daily (Placebo Comparator): Placebo orodispersible tablet twice daily
  Interventions: Drug: Placebo orodispersible tablet twice daily

INTERVENTIONS:
Drug: Budesonide 0.5mg orodispersible tablet twice daily
  Other Names: BUL 0.5mg BID
  Arms: Budesonide 0.5mg orodispersible tablet twice daily
Drug: Budesonide 1mg orodispersible tablet twice daily
  Other Names: BUL 1mg BID
  Arms: Budesonide 1mg orodispersible tablet twice daily
Drug: Placebo orodispersible tablet twice daily
  Other Names: Placebo BID
  Arms: Placebo orodispersible tablet twice daily

SUMMARY:
The purpose of this study is to prove the superiority of a 48-weeks treatment with budesonide orodispersible tablets versus placebo for the maintenance of clinico-pathological remission in patients with eosinophilic esophagitis.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent,
* Male or female patients, 18 to 75 years of age,
* Confirmed clinico-pathological diagnosis of eosinophilic esophagitis (EoE) according to established diagnostic criteria
* Clinico-pathological remission of EoE,
* A documented trial with proton pump inhibitors (PPIs) in order to rule out PPI-responsive esophageal eosinophilia,
* Negative pregnancy test in females of childbearing potential at baseline visit.

Exclusion Criteria:

* Clinical and endoscopic signs of gastroesophageal reflux disease (GERD),
* History of abnormal results in case of an optionally performed pH-monitoring of the distal esophagus,
* Patients with PPI-responsive esophageal eosinophilia
* Achalasia, scleroderma esophagus, or systemic sclerosis,
* Other clinically evident causes than EoE for esophageal eosinophilia,
* Any concomitant esophageal disease and relevant gastro-intestinal disease (celiac disease, inflammatory bowel disease, oropharyngeal or esophageal bacterial, viral, or fungal infection [candida esophagitis]),
* Any relevant systemic disease (e.g., AIDS, active tuberculosis),
* If careful medical monitoring is not ensured: cardiovascular disease, diabetes mellitus, osteoporosis, active peptic ulcer disease, glaucoma, cataract, or infection,
* Liver cirrhosis or portal hypertension,
* History of cancer in the last five years,
* History of esophageal surgery at any time or of esophageal dilation procedures within the last 8 weeks prior to screening visit,
* Upper gastrointestinal bleeding within 8 weeks prior to baseline visit,
* Existing or intended pregnancy or breast-feeding.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 204 (Actual)
Dates: Start 2016-01-15 (Actual); Primary Completion 2018-11-28 (Actual); Study Completion 2020-12-11 (Actual)

PRIMARY OUTCOMES:
Rate of patients free of treatment failure after 48 weeks of treatment. | 48 weeks

SECONDARY OUTCOMES:
Rate of patients with histological relapse | 48 weeks
Rate of patients with clinical relapse | 48 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Ralph Mueller, PhD, Study Director — Dr. Falk Pharma GmbH
Locations (1):
- Center for Digestive Diseases Eppendorf, Hamburg, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Biedermann L, Schlag C, Straumann A, Lucendo AJ, Miehlke S, Vieth M, Santander C, Ciriza de Los Rios C, Schmocker C, Madisch A, Hruz P, Hayat J, von Arnim U, Bredenoord AJ, Schubert S, Halstead M, Pfurr S, Mueller R, Schoepfer AM, Attwood S; International EOS-2 Study Group. Efficacy and Safety of Budesonide Orodispersible Tablets for Eosinophilic Esophagitis up to 3 Years: An Open-Label Extension Study. Clin Gastroenterol Hepatol. 2025 Nov;23(12):2144-2154.e6. doi: 10.1016/j.cgh.2024.10.034. Epub 2024 Dec 16. PMID 39694205